CLINICAL TRIAL: NCT04123275
Title: DCD III Study: a Multicentre Prospective Study to Identify Parameters Predicting Time to Death in Controlled Circulatory Death (cDCD) Donors and Prospective Validation of Previous Derived Prediction Models on Time to Death.
Brief Title: Prediction on Time to Death in Potential Controlled Donation After Circulatory Death (cDCD) Donors (DCD III Study)
Acronym: DCDIII
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: nw 2014-36
Record Dates: First submitted 2019-03-18; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-03

CONDITIONS: Tissue and Organ Procurement
Keywords: Validation studies; Withholding treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention wil be done. Patient characteristics and the standard care before and after withdrawal of life-sustaining treatment in all potential cDCD donors, will be studied. .

SUMMARY:
A considerable number of potential cDCD donors do not convert into actual organ donors because circulatory arrest does not occur within the predefined timeframe of warm ischemia after withdrawal of life-sustaining treatment. The main objective of this study is to determine parameters predicting time to death in potential cDCD patients.

DETAILED DESCRIPTION:
Controlled donation after circulatory death (cDCD) is a major source of organs for transplantation. Even though there is a well-established cDCD program in the Netherlands, there is still a considerable number of potential donors not being converted into actual organ donors. A potential cDCD donor poses considerable challenges in terms of a) identification of those dying within the predefined timeframe of warm ischemia, after withdrawal of life-sustaining treatment to circulatory arrest, b) managing them appropriately within the framework and resources of the intensive care unit, c) dealing with family expectations especially when failure to donation occurs, and d) efficient utilization of the organ procurement teams.

Factors associated with early circulatory collapse after treatment withdrawal include a younger age, non-triggered modes of artificial ventilation, high FiO2, the use of inotropes, and a low arterial pH. Another important factor which could influence the donor potential is end-of-life treatment. The practice of withdrawal of life support treatment (WLST) is highly variable between ICU's and countries. This influences the dying process and can thus have a large influence on the onset of cardio respiratory arrest. There is also wide variation in the use and dosage of additional sedation and analgesia during WLST and controversy exists regarding hastening or slowing down death.

Several attempts have been made to develop models to predict the time between treatment withdrawal and circulatory arrest, as this is crucial to a) proceed with organ donation, and b) the quality of the harvested organs. The selected patients however, where not always restricted to potential candidates for cDCD organ donation as patients with cancer and severe infection were also included.

Objective: Objectives of this study are: a) To determine parameters predicting time to death in potential cDCD patients b) To validate and update previous predicting models on time to death after withdrawal of life-sustaining treatment. c) To assess variation in withdrawal of life-sustaining treatment in the Netherlands and its influence on post mortal organ donor potential and actual post mortal organ donors.

Design and setting: Multicenter, observational, prospective cohort study of all potential cDCD patients of 3 university and 3 teaching hospitals in the Netherlands with diverse focus of attention

Methods: All potential cDCD patients participating in the cDCD protocol as defined by the Dutch Transplant Foundation admitted at the Intensive Care unit, will be included.

Participants: Mechanically ventilated ICU patients aged between 18 to 75 years. Brain dead patients will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients
* aged between 18 and 75 years old, where further treatment is futile.
* patients should meet the criteria of potential cDCD donors as defined by the Dutch Transplant Foundation

Exclusion Criteria:

* non-intubated patients
* younger than 18 years old
* brain dead patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All mechanically ventilated patients admitted at the Intensive Care Unit, aged between 18 and 75 years old who are eligible to enter the organ procurement protocol of the Dutch Transplant Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Duration (in minutes) on time to circulatory death after withdrawal of life-sustaining treatment, in cDCD patients | 36 months
  Development of a prediction tool to detect time to circulatory death (in minutes) in controlled donation after circulatory death patients (cDCD)

SECONDARY OUTCOMES:
Incidence of circulatory death in 60 minutes | 36 months
  Number of patients with circulatory death within 60 minutes
Incidence of circulatory death in 120 and 180 minutes | 36 months
  Number of patients when circulatory death occurs within the timeframe of 120 and 180 minutes
Doses analgesia | 36 months
  Doses analgesia provided before and during withdrawal of life support in milligrams per hour
Doses sedation | 36 months
  Doses sedation provided before and during withdrawal of life support in milligrams per hour
Incidence of withdrawal of endotracheal tube | 36 months
  Number of endotracheal tubes removed

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - ETZ, Tilburg
  - Isala clinics, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotsopoulos A, Vos P, Witjes M, Volbeda M, Franke H, Epker J, Sonneveld H, Simons K, Bronkhorst E, Mullers R, Jansen N, van der Hoeven H, Abdo WF. Prospective Multicenter Observational Cohort Study on Time to Death in Potential Controlled Donation After Circulatory Death Donors-Development and External Validation of Prediction Models: The DCD III Study. Transplantation. 2022 Sep 1;106(9):1844-1851. doi: 10.1097/TP.0000000000004106. Epub 2022 Mar 8. PMID 35266926
- [Derived] Kotsopoulos AMM, Vos P, Jansen NE, Bronkhorst EM, van der Hoeven JG, Abdo WF. Prediction Model for Timing of Death in Potential Donors After Circulatory Death (DCD III): Protocol for a Multicenter Prospective Observational Cohort Study. JMIR Res Protoc. 2020 Jun 23;9(6):e16733. doi: 10.2196/16733. PMID 32459638